CLINICAL TRIAL: NCT03696121
Title: Desmopressin for Reversal of Antiplatelet Drugs in Stroke Due to Haemorrhage (DASH)
Brief Title: Desmopressin for Reversal of Antiplatelet Drugs in Stroke Due to Haemorrhage
Acronym: DASH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 18040
Record Dates: First submitted 2018-06-08; First posted 2018-10-04 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Stroke, Acute
Keywords: intracerebral haemorrhage
MeSH Terms: conditions — Stroke; Cerebral Hemorrhage | interventions — Deamino Arginine Vasopressin; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Desmopressin injection
  Interventions: Drug: Desmopressin Injection
- Control (Placebo Comparator): Normal Saline
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Desmopressin Injection — Single dose 20 micrograms in 50ml Normal Saline as intravenous injection infused over 20 minutes
  Arms: Intervention
Drug: Normal saline — Single dose 50ml Normal Saline as intravenous injection infused over 20 minutes
  Arms: Control

SUMMARY:
Haemorrhagic stroke, an emergency caused by bleeding in the brain, often leads to death or long-term disability. A quarter of these patients are taking blood-thinning drugs (antiplatelet drugs, such as aspirin) because they are at risk of a heart attack or ischaemic stroke. Patients taking these drugs are more likely to die or be disabled if they have a haemorrhagic stroke. At present, there is no effective treatment for reversing their effects. Desmopressin is a drug which may reverse the effects of antiplatelet drugs and stop bleeding. The investigators would like to run a large randomised trial to see if Desmopressin can reduce the number of people who die or are disabled after haemorrhagic stroke.

DETAILED DESCRIPTION:
Intracerebral haemorrhage is a medical emergency, caused by a blood vessel bleeding directly into the brain. Outcome is directly related to the amount of bleeding that occurs. Many patients die early and others are left with significant disability. A quarter of all people with intracerebral haemorrhage are taking an antiplatelet drug, which is associated with larger volumes of brain haemorrhage and significantly worse outcomes. Four to five million people are taking antiplatelet drugs in the UK and use continues to rise in an ageing population.

Despite advances in treatment of ischaemic stroke, there is no effective drug treatment for intracerebral haemorrhage. Treatment for intracerebral haemorrhage has been identified as a priority area by Stroke Association and stroke survivors.

Desmopressin is a drug that reverses blood thinning effects of antiplatelet drugs, by indirectly increasing platelet adhesion, which the investigators hypothesise will minimise the devastating consequences of intracerebral haemorrhage associated with antiplatelet drugs. Desmopressin is commonly used in patients with inherited platelet dysfunction disorders and is an appealing treatment for antiplatelet-associated intracerebral haemorrhage. A recent systematic review did not find any randomised controlled trials evaluating desmopressin for antiplatelet-associated intracerebral haemorrhage. Desmopressin is affordable, available and could be implemented clinically across the UK and worldwide in the next five years with immediate benefit for stroke patients, their families and society.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years)
* Confirmed intracerebral haemorrhage on imaging
* Less than 24 hours from onset of symptoms [or from when last seen free of stroke symptoms]
* Prescribed and thought to be taking a daily oral antiplatelet drug in the preceding seven days (cyclooxygenase inhibitors, phosphodiesterase inhibitors or P2Y12 inhibitors)
* Signed consent (or waiver of consent).

Exclusion Criteria:

* Aneurysmal subarachnoid haemorrhage known at time of enrolment
* Haemorrhage suspected to be due to transformation of ischaemic stroke
* Haemorrhage known to be due to thrombolytic drug
* Haemorrhage known to be due to venous thrombosis
* Risk/s of fluid retention associated with desmopressin judged clinically significant by the attending physician (for example patients with pulmonary oedema and/or cardiac failure) - - Significant hypotension (systolic blood pressure <90mmHg)
* Known drug-eluting coronary artery stent in previous three months
* Allergy to desmopressin
* Pregnant or breast-feeding
* Life expectancy less than four hours, or planned for palliative care only
* Glasgow coma scale less than 5, mRS >4.

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Number of eligible patients who received allocated treatment | 90 days
  Number - higher number indicates feasibility of trial
Rate of eligible patients randomised | 18 months
  Shorter period of time to recruit number of patients indicates trial is feasibility;e
Proportion of eligible patients and randomised | 18 months
  Are there sufficient numbers of patients to justify a larger trial
Proportion of participants followed up at 90 days | 90 days
  Higher number indicates feasibility
Proportion of patients with full outcome data available, and reasons for non-availability | 90 days
  Higher number indicates feasibility
Proportion of eligible patients approached | 18 months
  Higher number indicates feasibility
Adherence to intervention | 18 months
  Higher number indicates feasibility

SECONDARY OUTCOMES:
Death or dependency at 90 days | 18 months
  Lower number indicates positive outcome
Number of patients dead or suffered serious adverse events | Day 28 and 90
  Number - higher number indicates worse outcome
Change in intracerebral haemorrhage volume at 24 hours | 24 hours
  Higher volume indicates worse outcome
Disability - Barthel index | Day 90
  Scores range from 0 - 100, with lower scores indicating increased disability.
Quality of life - EuroQol | Day 90
  Consists of two parts: a descriptive system (Part I) and a visual analogue scale (VAS) (Part II).
  Part 1 consists of 5 single-item dimensions. Scores range from 5 - 15 with lower scores indicating no problems to higher scores indicating extreme problems.
  Part II uses a vertical graduated VAS (thermometer) to measure health status, ranging from worst imaginable health state (0) to best imaginable health state (100).
Cognition - telephone MMSE | Day 90
  Scores are out of 22, with lower scores indicating cognitive impairment
Length of hospital stay | Day 90
  Number of days - higher number indicates longer length of stay
Discharge destination | 18 months
  Destination of participant following discharge from hospital
Health Economic assessment (EQ5D) | 90 Days
  Range 0-100, Higher score indicates better health
Serious adverse events (including thromboembolic events) | Day 90
  Higher volume indicates worse outcome
Change in factor vIII, Von Willebrand Factor antigen and Von Willebrand Factor activity will be assessed | One hour post administration of Desmopressin

CONTACTS AND LOCATIONS:
Overall Officials: Nikola Sprigg, Principal Investigator — University of Nottingham
Locations (1):
- Nottingham City Hospital, Nottingham, Notts, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Eilertsen H, Menon CS, Law ZK, Chen C, Bath PM, Steiner T, Desborough MJ, Sandset EC, Sprigg N, Al-Shahi Salman R. Haemostatic therapies for stroke due to acute, spontaneous intracerebral haemorrhage. Cochrane Database Syst Rev. 2023 Oct 23;10(10):CD005951. doi: 10.1002/14651858.CD005951.pub5. PMID 37870112
- [Derived] Desborough MJR, Al-Shahi Salman R, Stanworth SJ, Havard D, Brennan PM, Dineen RA, Coats TJ, Hepburn T, Bath PM, Sprigg N. Desmopressin for reversal of Antiplatelet drugs in Stroke due to Haemorrhage (DASH): protocol for a phase II double-blind randomised controlled feasibility trial. BMJ Open. 2020 Nov 10;10(11):e037555. doi: 10.1136/bmjopen-2020-037555. PMID 33172941